CLINICAL TRIAL: NCT06151587
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Different Concentrations of QLM3004 in Delaying the Progression of Myopia in Children
Brief Title: A Phase 3 Clinical Study of QLM3004 in Delaying Myopia in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QLM3004-301
Record Dates: First submitted 2023-11-20; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- QLM3004 Concentration 1 (Experimental): Solution low dose
  Interventions: Drug: QLM3004 Concentration 1
- QLM3004 Concentration 2 (Experimental): Solution medium dose
  Interventions: Drug: QLM3004 Concentration 2
- QLM3004 Concentration 3 (Experimental): Solution high dose
  Interventions: Drug: QLM3004 Concentration 3
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: QLM3004 Concentration 1 — Low dose of QLM3004 Ophthalmic Solution
  1 drop in each eye at bedtime
  Arms: QLM3004 Concentration 1
Drug: QLM3004 Concentration 2 — Medium dose of QLM3004 Ophthalmic Solution
  1 drop in each eye at bedtime
  Arms: QLM3004 Concentration 2
Drug: QLM3004 Concentration 3 — High dose of QLM3004 Ophthalmic Solution
  1 drop in each eye at bedtime
  Arms: QLM3004 Concentration 3
Other: Placebo — Vehicle
  Other Names: Control
  Arms: Placebo

SUMMARY:
Efficacy and Safety Study of QLM3004 in Myopic Children

DETAILED DESCRIPTION:
The study was divided into 2 phases, with Stage 1 being the primary efficacy and safety confirmation phase and Stage 2 a post-withdrawal observation period.

Stage 1:To evaluate the safety and efficacy of 3 concentrations of QLM3004 compared to Vehicle (placebo)for slowing the progression of myopia in children over a 96-week treatment period.

Stage 2:subjects will enter Period 2 of the study, and Period 2 will be a post-withdrawal observation period, which will not serve as a validation basis for the efficacy and safety of QLM3004.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years
* Myopia -1.00D to -4.00D spherical equivalent (SE) in both eyes as measured by cycloplegic autorefraction.
* Astigmatism ≤1.50 D in both eyes.
* Anisometropia ≤1.50 D SE.
* Informed consent signed by the subjects and/or their legal representatives

Exclusion Criteria:

* Suffering from serious systemic diseases
* Any eye disease that affect vision or refractive error
* Current or prior history of manifest strabismus, amblyopia, or other ocular pathologic changes
* Acute inflammatory disease or active infection of the eye in either eye, or a history of chronic ocular inflammation or recurrent episodes of ocular inflammation
* Best corrected distance visual acuity in both eyes<4.9
* Abnormal intra-ocular pressure (>21 mmHg or difference between two eyes >5mmHg)
* Current or previous form of myopia control, including but not limited to drugs, orthokeratology, progressive addition lenses, bifocal lenses, etc.
* Systemic or topical use of medications within 3 months that interfere with efficacy evaluation (excluding optometry)
* Allergy or hypersensitivity to atropine, excipients, cyclopentolate or fluorescein sodium
* Participants for whom the clinical significance of ophthalmologic examination abnormalities indicate that one or both eyes are not suitable candidates for treatment based upon the Investigator's medical judgment
* Participation of the drug clinical trial within three month and the device clinical trial within one month
* Anticipated long-term use of ocular or systemic oral corticosteroids during the study period
* Any other condition not suitable for the study per investigator's judgement

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 735 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in spherical equivalent determined by cycloplegic autorefraction at week 96. | 96 week
  Effectiveness Evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No